CLINICAL TRIAL: NCT06513819
Title: HIV and Alcohol Research Center Focused on Polypharmacy (HARP) Pilot 2 (2nd HARP Pilot Intervention)
Acronym: HARP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000038204; 1P01AA029545-01 (NIH)
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hiv; Alcohol Drinking; Fall; Cannabis Use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol Drinking | interventions — Motivational Interviewing; Methods

STUDY DESIGN:
Intervention Model Description: The Veterans Aging Cohort Study (VACS)-HIV database of 30 thousand veterans will be utilized to recruit eligible participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacist lead intervention (Experimental): Clinical pharmacists will be trained by a team with expertise in behavioral and HIV clinical care, and participate in a 10-hour training course with coaching sessions offered over the course of the study to ensure effective and consistent performance. Pharmacists will be guided by a manual designed to provide and walk them through the necessary skills to perform the pilot intervention easily and effectively. The manual will provide background information, study goals, and describe the critical components of the IMB-MI model and the HARP pilot interventions. An easy to follow, step-by-step approach to performing the intervention will be included. The study protocol to be followed by the clinical pharmacists will be included in the manual along with additional motivational and troubleshooting strategies. Systematic feedback regarding intervention fidelity will be provided by the Evaluation Team.
  Interventions: Behavioral: Information Motivation Behavioral and Motivational Interviewing (IMB-MI) technique

INTERVENTIONS:
Behavioral: Information Motivation Behavioral and Motivational Interviewing (IMB-MI) technique — Delivered by a clinical pharmacist who will employ IMB-MI in informational, participant-centered discussions in which the clinical pharmacist and the participant collaboratively discuss the harms of alcohol use (with or without concurrent use of cannabis) and polypharmacy (specifically neurocognitively active medications), the relationship of these exposures to fall risk and NCEs, and how to mitigate these harms. Together pharmacist and participant will develop a plan for change in alcohol and polypharmacy use, self-monitoring, medications of concern, symptoms, and any additional resources needed. The goal of the intervention being to help patients stop or decrease alcohol use and stop medications in situations where it is safe to do so and agreed upon by the primary provider (but substitutions will be made if necessary).

SUMMARY:
The focus of this pilot will be on falls and neurocognitive symptoms, and the impact of alcohol, cannabis use, and medications on these outcomes. The rationale is that alcohol use at any level may interact with neurocognitively active medications, alcohol, and cannabis use leading to falls and impaired cognition.

DETAILED DESCRIPTION:
Pilot 2 will consist of a brief pharmacist-led intervention for patients with HIV who consumed alcohol in the past month, take 5 or more medications in addition to their antiretroviral therapy (ART) regimen, and one or more of their non ART medications is known to have neurocognitive effects (NCEs, not including antiseizure medications).

Prior to starting intervention: The study staff will recruit and obtain consent. Those who do not opt-out of the study will be contacted by phone and study staff will verify the individual currently consumes alcohol, administer the Alcohol Symptom Checklist, obtain verbal consent for the study, and verify their contact information. The Alcohol Symptom Checklist will be given as a screen during this first contact to determine level of alcohol use. Study staff will inform the participant about the self-administered blood spot test for phosphatidylethanol (PEth) and subsequently send a video with step-by-step instructions on how to perform these tests in a text message after the call. Finally, staff will schedule a brief call (estimated time of 15-20 minutes) with a VA clinical pharmacist assisting with recruitment approximately 3-5 days ahead to conduct a medication reconciliation. After enrollment is complete, a study staff member will request that a home test kit for PEth and the initial survey be sent to the participant from the West Haven Coordinating Center. Once completed, the participant will be asked to put the questionnaire in the self-addressed, stamped envelope and mail it back to the West Haven Coordinating Center. A separate envelope will be provided to send the biomarker samples directly to the analytic lab, processed at the United States Drug Testing Laboratories (USDTL) for rapid analysis.

After enrollment, participants will be contacted by a designated VA clinical pharmacist 1-2 days after the recruitment phone call to confirm a reconciliation of the participant's list of current medications. At this time, the clinical pharmacist will also schedule the intervention call that will take place four weeks ahead.

The intervention will be conducted by an additional group of VA clinical pharmacists specifically trained in IMB-MI procedures prior to the start of the study, following a training plan developed and delivered by expert advisors in the Risk Communication Resource Core of HARP, and trained to criterion standard. This training approach has been successfully used in our previous studies. The intervention will be digitally recorded to allow us to monitor fidelity. These recordings will be stored on our servers behind the VA firewall. Only those who are monitoring intervention fidelity will have access to these recordings.

4 weeks following the intervention call, the clinical pharmacist will check-in with the participant and inquire about their chosen goals and the progress they may or may not have been making, along with motivators and/or setbacks. The clinical pharmacists will remind the participant to complete the immediate post intervention survey (information, motivation, behavioral skills, importance and confidence, behavioral intentions ~5 minutes) once it arrives, and to return it in the enclosed postage paid. The participant is to mail the survey, along with completed monitoring forms from the previous weeks, back to the West Haven Coordinating Center in the self-addressed, stamped envelope provided.

6 months after the interview, participants will be sent a second PEth home test kit to measure changes in alcohol consumption with return envelope, along with a final 6-Month Post Intervention Survey measuring the items listed above, along with feedback questions related to feasibility of the study, clarity of instructions and provided information, PEth test, and open-ended questions for the participant to write in their own comments. We will also check VA EHR pharmacy data.

Finally, we will recontact a subset of participants for qualitative interviews that will elicit their feedback on the intervention. This information includes but is not limited to asking how difficult they found self-administering the PEth test, assessing whether their personalized risk estimate influenced their thinking on their alcohol or medication use, their views on cannabis use, their views on how clearly the clinical pharmacists were able to communicate risk information, how well they liked receiving the intervention from a clinical pharmacist, and the usefulness of the intervention provided to reduce alcohol use. These interviews will be targeted to occur within one week after the 30-day follow-up, but we will allow up to 1 month. We will conduct these interviews by telephone or Microsoft Teams. These conversations will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* have visited a local VA site in within the past year
* had an AUDIT-C indicating current alcohol use
* taking 5 or more non-ART medications, including an NCAM (i.e., benzodiazepines, opioids, muscle relaxants, sleeping medication, and selective serotonin reuptake inhibitors)

Exclusion Criteria:

* Inpatient individuals
* Patients with an Alcohol Use Disorder (AUD) diagnosis in the past 12 months
* Patients who test positive on the Alcohol Symptom Checklist for moderate or severe AUD during the screening process

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Ability to meet enrollment target of 100 participants | Week -2 to Week 0
  Enrollment of 100 Participants: Week -2: Gather list of 100 eligible patients from the online VACS-HIV Index database; Send opt-out letter with study information and contact number. Week -2 to Week 0: Track patients for 2 weeks and note which have opted out. Week 0: Contact patients who have not opted-out; enroll, screen, and conduct medication reconciliation phone call; Send out pre-intervention package.
Feasibility: Ability to deliver the complete intervention | Week 3 and week 7
  Week 3: 1-hour intervention call between VA clinical pharmacist and participant Week 7: 30-minute booster call between VA clinical pharmacist and participant
Feasibility:Percentage of Completion of Study Items | up to Month 9
  Percentage of completion of study items (Pre-Intervention Survey, Phosphatidylethanol Test, Post-Intervention Survey, 6-Month Post Intervention Survey, Phosphatidylethanol Test 2). Higher percentage indicates more completion of study items.
Acceptability: comfort, comprehensibility/helpfulness of content | Week 7, Month 9 and Month 9,Week 3
  Assessed using a series of multiple-choice feedback and open-ended questions on Post-Intervention Survey and 6-Month Post Intervention Survey and a series of prompts on final semi-structured interview focused on feedback from participant
Acceptability: acceptability of PEth tests | Week 7, Month 9 and Month 9,Week 3
  Assessed using a series of multiple-choice feedback and open-ended questions on Post-Intervention Survey and 6-Month Post Intervention Survey and a series of prompts on final semi-structured interview focused on feedback from participant

SECONDARY OUTCOMES:
Neurocognitive symptoms mean score | Weeks 0, 7 and Month 9
  Participants will answer 10 questions asking on a 4 point scale of "no or less" to "lot more" difficulty with different everyday cognitive responsibilities such as losing track of a current task, difficulty remembering appointments, etc. compared to 5 years ago, 4 weeks ago and 6 months ago. Total score range from 0-30. Higher scores will indicate higher cognitive dysfunction, and lower scores will indicate clearer cognitive function.
Fall Risk | Weeks 0, 7 and Month 9
  Participants will be asked about their history of falls and fractures to observe the interaction between cognitive decline and frequency of falls.The predicted probability of a fall is: Phat = 1/ (1 + exponent^(-Linear Predictor)
Readiness to Change mean score | Weeks 0, 7 and Month 9
  A series of 6 questions asking participants on a Likert scale of 1= not at all to 10=extremely regarding their readiness, confidence and importance related to change behaviors about alcohol (3 questions) and medications (3 questions). Total score range 6-60. Higher scores will indicate a strong readiness to change.
Alcohol Use assessed using PEth | Weeks 0 and Month 9
  Participants will complete 2 fingerstick blood spot phosphatidylethanol (PEth) tests on their own at home using items the study staff will provide in the mail. PEth testing uses blood to measure alcohol use by detecting direct alcohol biomarkers in the bloodstream. A positive test with a score <8 indicates alcohol use. Score: <8 = Negative, 8-20 = Low to moderate alcohol use, 20-50 = Heavy alcohol use, 50> = Very heavy alcohol use
Alcohol Use Survey mean score | Weeks 0, 7 and Month 9
  Participants will answer a series of questions on a 4-point scale of "Strongly Disagree" to "Strong Agree" related to their alcohol use. Each question is scored on a scale of 0 to 4, with a total possible score ranging from 0 to 40. Higher scores indicate a greater likelihood of alcohol-related problems or AUD.
Cannabis Use | Weeks 0, 7 and Month 9
  1 question asking participants about cannabis use, Yes/No.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Justice, MD, PhD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No